CLINICAL TRIAL: NCT05052749
Title: Effects of High Intensity Resistance Training in Postmenopausal Women
Brief Title: High Intensity Resistance Training In Postmenopausal Women (HIRT)
Acronym: HIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00915 Qurat-ul-Ain
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Post Menopause

STUDY DESIGN:
Intervention Model Description: This will be a single factor, Pretest-Posttest Control Group Design with parallel assignment of patients in to two groups.
Who Masked: Participant
Masking Description: Female participants in clinical trial will be kept blind about their exercise group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Resistance Training (HIRT) (Experimental): In this HIRT group, participants will perform warm-up activity for 15 minutes then high intensity resistance exercises with 120 seconds of rest interval between each set of exercise and between exercises respectively. After that, generalized stretching exercises as a cool down activity will be performed by the participants. Participants will perform exercises twice weekly, 40-50 minutes/session for 12 weeks under supervision.
  Interventions: Other: High Intensity Resistance Training (HIRT)
- Low-moderate Resistance Exercise Training (Active Comparator): In this low-moderate resistance training group, participants will perform warm-up activity for 15 minutes then low-moderate intensity resistance exercises with 120 seconds of rest interval between each set of exercise and between exercises respectively. After that, generalized stretching exercises as a cool down activity will be performed by the participants. Participants will perform exercises twice weekly, 40-50 minutes/session for 12 weeks under supervision.
  Interventions: Other: Low-moderate Resistance Exercise Training

INTERVENTIONS:
Other: High Intensity Resistance Training (HIRT) — High Intensity Resistance Exercises Supervised High Intensity Resistance Training with 15 minutes of cycling as a warm-up activity then HIRT through Quadriceps drill, Squats, Lunges, Leg press, Biceps curls and Deadlift with 120 seconds of rest interval between each set of exercise and between exercises will be performed by the participants with appropriate cool down through generalized stretching exercises. Participants will perform exercises twice weekly, 40-50 minutes/session for 12 weeks respectively.
  Arms: High Intensity Resistance Training (HIRT)
Other: Low-moderate Resistance Exercise Training — Supervised Low-moderate Resistance Training with 15 minutes of cycling as a warm-up activity then Quadriceps drill, Squats, Lunges, Leg press, Biceps curls and Deadlift with 120 seconds of rest interval between each set of exercise and between exercises will be performed by the participants with appropriate cool down through generalized stretching exercises. Participants will perform exercises twice weekly, 40-50 minutes/session for 12 weeks respectively.
  Arms: Low-moderate Resistance Exercise Training

SUMMARY:
Menopause is defined as a permanent cessation of menstrual cycle for 12 months due to intrinsic diminution of ovarian oocytes among women in older age. Globally reported mean age for menopause is 48.78 years (ranges from 46-52 years). Menopausal age reported among Asian and African population was lower as compared to European women . Among postmenopausal women, age related various central nervous system, musculoskeletal, urogenital, metabolic and skin changes ensue along with osteoporosis (T-score = ≤ -2.5) and decreased bone mineral density due to estrogen deficiency that is directly associated with fragility fractures and disability among this age group. Therefore, recruitment of older adults in resistance training program is crucial in inducing increases in muscle strength and ameliorating glucose tolerance and increased insulin sensitivity along with improvements in BMD and BMR.

DETAILED DESCRIPTION:
Physical activity is extremely crucial in maintaining quality of life and estrogen metabolism among postmenopausal women, owing to the increased risk of falls, age related decline in cardiopulmonary, musculoskeletal endurance and cognitive capacity. In Pakistan, fitness of women specifically of postmenopausal age group is ignored due to some cultural norms. Performance of physical activity in the form of resistance training (RT) is one of the best known methods to improve physical fitness in the elderly. So the current study is planned with objectives to determine effects of High Intensity Resistance Training in Postmenopausal Women. Supervised exercise training will be provided for 3 months and functional performance will be measured accordingly.

After initial screening of postmenopausal women including history and anthropometric details, females meeting inclusion criteria and willing to participate in high intensity resistance exercise trial will be recruited in the study. After that; physical fitness, performance base testing for functional performance outcome measures and MENQOL assessment will be done at baseline and after 3 months. Patients will perform resistance training twice a week, 40-50 min/session for 12 weeks respectively. It is hypothesized that supervised high intensity resistance training will improve functional performance, physical fitness and Quality of life among postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Age: 45-70 years
* Sedentary life style

Exclusion Criteria:

* High risk of fracture as calculated by WHO online FRAX tool.
* Presence/history of fragility fracture.
* MMSE < 20
* Systemic illness: hyperthyroidism, hyperparathyroidism, renal failure, any malignancy, extensive radiation exposure.
* Any orthopedic injury/disorder hindering performance of exercise.
* Not willing for exercise.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
10RM leg press | 3 months
  Assessed from baseline. 10 RM is used to assess maximum muscle strength that is to extend knee 10 times against maximum resistance. Weight will be recorded in Kgs.
  [Time Frame: 3 Months]
10RM dead lift (kg) | 3 months
  Assessed from baseline. 10 RM is used to assess maximum muscle strength that is to lift weight 10 times against maximum resistance. Weight will be recorded in Kgs.
Sit and reach test (cm) | 3 months
  Assessed from baseline. It is linear flexibility test used to measure extensibility of hamstrings and lower back. Participant will perform test in seated position with extended knees, distance between extended fingers and top of the toe will be recorded in cm.
Sit and stand test (reps) | 3 months
  Assessed from baseline. In this test participant will rise to full standing position from seated position without using armrests of chair and researcher will count the number of complete stand from sitting position within 30 seconds. Inaccurately accomplished stands will not be counted.
Plank test (sec) | 3 months
  Assessed from baseline. It is fitness test that measures the endurance of core stabilizing muscles. Participants will be in prone position with elbow flexion at 90° and forearm resting on floor and toes touching the floor. Two trials will be recorded with 1.5 minutes of rest interval between attempts and extensive isometric time will be used for analysis.
6 - minutes' walk test (sec) | 3 months
  Assessed from baseline. It is sub-maximal exercise test used to evaluate aerobic capacity and endurance. Participant will walk in 30-metre walkway with marked ends for 6 minutes. Patient will be permitted to slow down, stop or rest when required. Record the distance walked in 6 minutes' duration with vital signs monitoring.
Gait speed | 3 months
  Assessed from baseline. Gait speed test is used to assess functional mobility of an individual. Gait speed will be measured from 6-m distance in 10-m track using stopwatch with 2 meters for acceleration and 2 meters for deceleration respectively. Two trials will be performed and then average score will be taken for analysis. Participant will start walking with dominant foot with maximum pace possible.
Menopause specific Quality of life (MENQOL) | 3 months
  Assessed from baseline. Menopause specific Quality of life is the tool used to assess quality of life among postmenopausal women in the past month. It has four domains of menopausal symptoms; vasomotor, psychosocial, physical and sexual. A total of 29 items in a 6 point Likert-scale is used, with 0 means not at all bothered and 6 means extremely bothered. the minimum score is 0 and maximum is 174.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, RCRAHS Westridge campus, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu D, Chung HF, Dobson AJ, Pandeya N, Giles GG, Bruinsma F, Brunner EJ, Kuh D, Hardy R, Avis NE, Gold EB, Derby CA, Matthews KA, Cade JE, Greenwood DC, Demakakos P, Brown DE, Sievert LL, Anderson D, Hayashi K, Lee JS, Mizunuma H, Tillin T, Simonsen MK, Adami HO, Weiderpass E, Mishra GD. Age at natural menopause and risk of incident cardiovascular disease: a pooled analysis of individual patient data. Lancet Public Health. 2019 Nov;4(11):e553-e564. doi: 10.1016/S2468-2667(19)30155-0. Epub 2019 Oct 3. PMID 31588031
- [Background] Monteleone P, Mascagni G, Giannini A, Genazzani AR, Simoncini T. Symptoms of menopause - global prevalence, physiology and implications. Nat Rev Endocrinol. 2018 Apr;14(4):199-215. doi: 10.1038/nrendo.2017.180. Epub 2018 Feb 2. PMID 29393299
- [Background] Maillard F, Rousset S, Pereira B, Traore A, de Pradel Del Amaze P, Boirie Y, Duclos M, Boisseau N. High-intensity interval training reduces abdominal fat mass in postmenopausal women with type 2 diabetes. Diabetes Metab. 2016 Dec;42(6):433-441. doi: 10.1016/j.diabet.2016.07.031. Epub 2016 Aug 24. PMID 27567125
- [Background] Daly RM, Dalla Via J, Duckham RL, Fraser SF, Helge EW. Exercise for the prevention of osteoporosis in postmenopausal women: an evidence-based guide to the optimal prescription. Braz J Phys Ther. 2019 Mar-Apr;23(2):170-180. doi: 10.1016/j.bjpt.2018.11.011. Epub 2018 Nov 22. PMID 30503353
- [Background] Socha M, Fraczak P, Jonak W, Sobiech KA. Effect of resistance training with elements of stretching on body composition and quality of life in postmenopausal women. Prz Menopauzalny. 2016 Mar;15(1):26-31. doi: 10.5114/pm.2016.58770. Epub 2016 Mar 29. PMID 27095955
- [Background] Dias RKN, Penna EM, Noronha ASN, de Azevedo ABC, Barbalho M, Gentil PV, Coswig VS. Cluster-sets resistance training induce similar functional and strength improvements than the traditional method in postmenopausal and elderly women. Exp Gerontol. 2020 Sep;138:111011. doi: 10.1016/j.exger.2020.111011. Epub 2020 Jun 24. PMID 32592830